CLINICAL TRIAL: NCT01723930
Title: Transpulmonary Gradient of Inflammation Biomarkers and Pulmonary Vascular Resistance in Acute Respiratory Failure After Cardiac Surgery Under Cardiopulmonary Bypass
Brief Title: Transpulmonary Gradient After Cardiac Surgery Under Cardiopulmonary Bypass
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 5328
Record Dates: First submitted 2012-11-06; First posted 2012-11-08 (Estimated); Last update posted 2012-11-08 (Estimated); Status verified 2012-11

CONDITIONS: Acute Respiratory Distress Syndrome After Cardiac Surgery Under Cardiopulmonary Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Get a better understanding of the pathophysiological processes of acute respiratory failure following cardiopulmonary bypass to initiate timely therapies targeted on a cell line.

Demonstrate that there is a relationship between increased transpulmonary gradients of inflammation biomarkers (sRAGE, sICAM-1, SPB, PAI-1, ROS) and pulmonary vascular resistance on the one hand and alveolo-capillary gas exchange on the other hand after cardiac surgery under cardiopulmonary bypass.

ELIGIBILITY:
Inclusion Criteria:

* Patient man or woman > 18 y.o.
* Patient has signed informed consent prior to the study
* Patient affiliated to a social security administration
* Patient operated on for cardiac surgery at the University Hospital of Strasbourg.
* Patient at high risk for postoperative respiratory failure defined by a SLIP score (Kor et al.) ≥ 22 Kor:

  * High-risk cardiac intervention under cardiopulmonary bypass (19 pts)
  * COPD (10 pts)
  * Diabetes (6 pts)
  * gastroesophageal reflux (7 pts)
  * Alcohol abuse (11 pts)
* Scheduled use of a pulmonary artery catheter and a left atrial catheter

Exclusion Criteria:

* Inability to obtain informed consent from the patient and / or unable to give informed patient information (difficulty understanding ...)
* Urgent surgery (<24h)
* Acute heart failure
* Patient ventilated preoperatively
* Allergy to Latex
* Persons deprived of liberty or under judicial protection
* Patient placed under guardianship
* Pregnancy
* Breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recruitment concerns only patients with high risk of postoperative respiratory failure (SLIP score > 22).
Sampling Method: Non-Probability Sample
Enrollment: 30

PRIMARY OUTCOMES:
transpulmonary gradients of inflammation biomarkers (sRAGE, sICAM-1, SPB, PAI-1, ROS) and pulmonary vascular resistance | during the surgery
  Demonstrate that there is a relationship between increased transpulmonary gradients of inflammation biomarkers (sRAGE, sICAM-1, SPB, PAI-1, ROS) and pulmonary vascular resistance on the one hand and alveolo-capillary gas exchange on the other hand after cardiac surgery under cardiopulmonary bypass.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Strasbourg, Alsace, France